CLINICAL TRIAL: NCT02163668
Title: Effects of an 8-month Yoga Intervention on Bone Metabolism in Healthy Middle-aged Premenopausal Women: A Randomized Controlled Study
Brief Title: Effects of Yoga on Bone Metabolism in Premenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Principal Investigator, Debra Bemben, Professor, University of Oklahoma
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OUYogaStudy
Record Dates: First submitted 2014-06-09; First posted 2014-06-16 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-06

CONDITIONS: Bone Health; Osteoporosis
Keywords: Yoga; Bone turnover markers; Bone strength; Bone mineral density
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yoga group (Experimental): 8 months of progressive Yoga training
  Interventions: Other: Yoga Group
- Control group (No Intervention): No training, just pre and post testing

INTERVENTIONS:
Other: Yoga Group — 8 months of Yoga training
  Arms: Yoga group

SUMMARY:
This study examined the effects of 8 months of Yoga training on bone density and bone turnover markers in premenopausal women, ages 35-50 years. The style of Yoga used was power Yoga that involved postures with a jumping component. The investigators hypothesized that the Yoga intervention would result in beneficial improvements in bone turnover markers, by increasing the bone formation marker and decreasing the bone resorption marker.

ELIGIBILITY:
Inclusion Criteria:

* participants had not been engaged in resistance training or in Yoga exercise for at least 12 months prior to the study
* did not have chronic back or joint problems or cardiovascular disease
* not taking antihypertensive drugs or any medication that affects bone density
* not taking hormonal contraception
* they self-reported having regular menstrual cycles.

Exclusion Criteria:

* body weight more than 300 pounds

Ages: 35 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2009-09; Primary Completion 2010-06 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Change in bone mineral density from baseline to 8 months | pre and post 8 months training
change in bone turnover markers | pre and post 8 month intervention
change in tibia bone characteristics | pre and post 8 month intervention
  changes in volumetric bone mineral density and bone strength of the non-dominant tibia assessed by peripheral Quantitative Computed Tomography (pQCT)
Changes in muscular strength | pre and post 9 month intervention
  Isotonic 1 repetition maximum (1RM) for 4 lower body and 2 upper body resistance exercises
Change in arterial compliance | pre and post 8 month interventon
  Arterial compliance of the large and small arteries was assessed using Pulse Contour analysis.
Change in Insulin-like Growth Factor-1 (IGF-I) and Insulin-like Growth Factor BP3 (IGFBP3) | pre and post 8 month intervention

SECONDARY OUTCOMES:
Daily Calcium intake | pre and post 8 month intervention
  Calcium intake is a potential confounding variable. Participants were encouraged to increase their calcium intakes if found to be low before the intervention began.
Menstrual History | pre and post 8 month intervention
  This information was used to monitor menstrual characteristics to ensure they were still premenopausal at the post test.
Dietary intake | At baseline at the same time as other outcomes, about 2 weeks before the beginning of the yoga training
  Three day dietary logs were recorded by participants before the exercise intervention. They were analyzed for caloric intake and nutrient composition using the Diet Analysis Plus 9 software.
Change in physical activity levels | pre and post 8 month intervention
  Physical activity levels estimated by the bone-specific physical activity (PA) questionnaire to monitor their PA outside of the intervention
Change in body composition | pre and post 8 month intervention

CONTACTS AND LOCATIONS:
Overall Officials: Debra A Bemben, PhD, Principal Investigator — Department of Health and Exercise Science, University of Oklahoma
Locations (1):
- Department of Health and Exercise Science, University of Oklahoma, Norman, Oklahoma, United States

REFERENCES:
- [Background] Phoosuwan M, Kritpet T, Yuktanandana P. The effects of weight bearing yoga training on the bone resorption markers of the postmenopausal women. J Med Assoc Thai. 2009 Sep;92 Suppl5:S102-8. PMID 19891384
- [Background] Chan K, Qin L, Lau M, Woo J, Au S, Choy W, Lee K, Lee S. A randomized, prospective study of the effects of Tai Chi Chun exercise on bone mineral density in postmenopausal women. Arch Phys Med Rehabil. 2004 May;85(5):717-22. doi: 10.1016/j.apmr.2003.08.091. PMID 15129394